CLINICAL TRIAL: NCT03199612
Title: The Role of Hemolysis in Promoting Thrombosis During Mechanical Circulatory Support With Continuous Flow Pumps (Aim 2)
Brief Title: Sildenafil To Prevent Clot
Acronym: SToPClot
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-7404; 5K23HL145140 (NIH)
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Thrombosis; Hemolysis
Keywords: Thrombosis during Continuous Flow Pump Support
MeSH Terms: conditions — Thrombosis; Hemolysis | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Placebo controlled randomized trial with 1:1 enrollment in each study arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sildenafil (Active Comparator): Baseline blood samples and study measurements will be acquired. Then 20 mg of the study drug will be administered. Then BP will be recorded every 30 minutes for two hours. If BP is stable (drop is < 5 mmHg after 2 hours and patient is asymptomatic), patient will proceed to take 20 mg of the study drug every 8 hours. The patient will return to clinic on day 8 and 20 mg of the study drug will be administered. After 2 hours blood samples and study measurements will be collected and the patient will resume 20 mg of the study for the next two doses. The patient will return for a third clinic visit on the next day and if BP is in the acceptable range, 40 mg of the study drug will be administered. If BP remains stable for 2 hours, then the patient will continue taking 40 mg every 8 hours. The patient will return to clinic on day 15 for a final study visit and will be given the last 40 mg dose of the study drug and after 2 hours blood samples and study measurements will be taken.
  Interventions: Drug: Sildenafil
- Placebo Oral Tablet (Placebo Comparator): Negative control to understand the potential changes in platelet activation and aggregation in comparison to sildenafil.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sildenafil — To conduct a randomized placebo controlled study to test the hypothesis that platelet activation and aggregation during ongoing low level hemolysis in outpatients on chronic CF pump support can be reduced by sildenafil.
  Other Names: Viagra; Revatio
  Arms: Sildenafil
Drug: Placebo Oral Tablet — Negative control to understand the potential changes in platelet activation adn aggregation in comparison to sildenafil.
  Other Names: Sildenafil matching placebo
  Arms: Placebo Oral Tablet

SUMMARY:
The advent of continuous flow (CF) pumps for patients with severe heart failure has led to marked improvements in survival; however, pump operation remains fraught with adverse thrombotic events. This climbing rate of thrombosis and stroke during CF pump support has led to a recent warning by the US Food and Drug Administration. Despite a rising incidence of pump thrombosis and its downstream complications of stroke, the hematologic mechanisms behind these devastating adverse events remain uncertain. Recently, it has been recognized that CF pump induced hemolysis precedes and is associated with thrombosis. In-vitro studies show increased platelet function with exposure to products of hemolysis, which is also known to occur in diseases of intravascular hemolysis such as sickle cell anemia. This proposal will investigate if hemolysis associated increased platelet function can be reduced by a potentiation of nitric oxide signaling by an oral phosphodiesterase-5 inhibitor, sildenafil. Elucidating mechanisms of hemolysis induced thrombosis may inform best strategies for prevention of end organ damage and maintaining optimal CF pump operation.

DETAILED DESCRIPTION:
Despite the remarkable improvements in survival with durable continuous flow (CF) pumps and the clear lifesaving effects of Impella and veno-arterial extracorporeal membrane oxygenation (VA ECMO), serious adverse hematological events such as bleeding and thrombosis create substantial morbidity and mortality and remain major barriers for further expansion of this technology. In particular, thrombosis is a devastating adverse event during CF pump support as it can lead to stroke, device stoppage, and hemodynamic collapse. Although the annual incidence of pump thrombosis has been reported to range from 8 to nearly 30%, the pathobiological mechanisms of thrombus formation during CF pump support with ongoing anticoagulation remain elusive. Our preliminary data associates hemolysis, which is inherent to such devices due to high shear stress, with subsequent formation of thrombosis and stroke, possibly through increasing platelet activation and aggregation. Our prelim data and drawing from a body of literature from diseases of intravascular hemolysis such as sickle cell anemia suggest that free hemoglobin released during hemolysis, which reduces NO levels, may be activating platelets. In retrospective analysis, we have noted a significant reduction in mean platelet volume (potential in-vivo marker of platelet activation), thrombosis and stroke with concurrent sildenafil administration. However, this mechanism and efficacy of NO signaling enhancers such as sildenafil remains to be proven during CF pump support.

Aim: To conduct a randomized placebo controlled study to test the hypothesis that platelet activation and aggregation, endothelial dysfunction and pro-thrombotic inflammation in outpatients on chronic CF pump support can be reduced by sildenafil.

ELIGIBILITY:
Inclusion:

-Adult outpatients (≥18 years old) with ongoing durable CF pump support.

Exclusion:

* Taking sildenafil or nitrates for clinical indications
* Ongoing infection
* Unwilling or unable to give written, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Saeed, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil: Baseline blood samples and study measurements will be acquired. Then 20 mg of the study drug will be administered. Then BP will be recorded every 30 minutes for two hours. If BP is stable (drop is < 5 mmHg after 2 hours and patient is asymptomatic), patient will proceed to take 20 mg of the study drug every 8 hours. The patient will return to clinic on day 8 and 20 mg of the study drug will be administered. After 2 hours blood samples and study measurements will be collected and the patient will resume 20 mg of the study for the next two doses. The patient will return for a third clinic visit on the next day and if BP is in the acceptable range, 40 mg of the study drug will be administered. If BP remains stable for 2 hours, then the patient will continue taking 40 mg every 8 hours. The patient will return to clinic on day 15 for a final study visit and will be given the last 40 mg dose of the study drug and after 2 hours blood samples and study measurements will be taken.
  Sildenafil: To conduct a randomized placebo controlled study to test the hypothesis that platelet activation and aggregation during ongoing low level hemolysis in outpatients on chronic continuous flow (CF) pump support can be reduced by sildenafil.
Period: Overall Study
Arm/Group | Sildenafil | Placebo Oral Tablet
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Oral Tablet: Negative control to understand the potential changes in platelet activation and aggregation in comparison to sildenafil.
  Placebo Oral Tablet: Negative control to understand the potential changes in platelet activation and aggregation in comparison to sildenafil.
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo Oral Tablet | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [45 to 63] | 56 [44 to 68] | 55 [44 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non Hispanic Black | 5 | 4 | 9
  Non Hispanic White | 1 | 3 | 4
  Hispanic | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Adenosine Diphosphate (ADP)
Description: During the study period platelet activation and aggregation will be measured from drawn blood samples. Platelet rich plasma will be isolated from these samples and platelet aggregometry will be used to measure platelet activation and aggregation. Platelet activation and aggregation is measured as an area under the curve (AUC) derived as the resistance (ohms) x time (s). There is no reference range for ADP induced AUC. Higher values of AUC indicate greater platelet aggregation.
Time Frame: Baseline, day 8 and day 15
Population: 1 participant in the sildenafil group was not able to tolerate 40 mg and did not reach the 15 day endpoint.
Measure: Median (Inter-Quartile Range); unit: omhs x seconds (AUC)
Arm/Group | Sildenafil | Placebo Oral Tablet
Number analyzed (Participants) | 10 | 10
omhs x seconds (AUC)
  Baseline | 50 [35 to 67] | 20 [4 to 35]
  Day 8 | 50 [25 to 60] | 6 [0.3 to 40]
  Day 15: number analyzed (Participants) | 9 | 10
  Day 15 | 38 [19 to 69] | 27 [2 to 60]

2. Secondary Outcome: Pro-thrombotic Inflammation as Measured by High-sensitivity C-reactive Protein (hs CRP)
Description: During the study period pro-thrombotic inflammatory markers, including hs CRP (mg/L) in serum will be measured by ELISA. The upper limit of normal reference for hs CRP is 0.5 mg/dL. Higher values of hs CRP indicate greater pro-thrombotic inflammation.
Time Frame: Baseline, day 8 and day 15
Population: 1 participant in the sildenafil group was not able to tolerate 40 mg and did not reach the 15 day endpoint.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Sildenafil | Placebo Oral Tablet
Number analyzed (Participants) | 10 | 10
mg/L
  Baseline | 2.2 [1.31 to 3.63] | 2.2 [1.0 to 3.1]
  Day 8 | 2.9 [1.75 to 4.05] | 2.20 [1.04 to 3.07]
  Day 15: number analyzed (Participants) | 9 | 10
  Day 15 | 2.57 [0.88 to 5.02] | 2.2 [0.75 to 3.98]

3. Secondary Outcome: Pro-thrombotic Inflammation as Measured by Fibrinogen
Description: During the study period pro-thrombotic inflammatory markers including fibrinogen (mg/dL) will be measured by ELISA. The upper limit of normal reference for fibrinogen is 187-502 mg/dl. Higher values of fibrinogen indicate greater thrombo-inflammation.
Time Frame: Baseline, day 8 and day 15
Population: 1 participant in the sildenafil group was not able to tolerate 40 mg and did not reach the 15 day endpoint.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Sildenafil | Placebo Oral Tablet
Number analyzed (Participants) | 10 | 10
mg/dl
  Baseline | 355 [313 to 388] | 334 [277 to 372]
  Day 8 | 392 [324 to 434] | 311 [295 to 345]
  Day 15: number analyzed (Participants) | 9 | 10
  Day 15 | 398 [324 to 440] | 345 [292 to 389]

4. Other Pre Specified Outcome: Serum Angiopoietin-2 to Angiopoietin-1 Ratio
Description: Mediator of vascular remodeling. This is a relative unit and there is no reference range in the context of magnetically levitated left ventricular assist device support. A higher Angiopoietin-2 to Angiopoietin-1 ratio indicates greater microvascular remodeling and inflammation.
Time Frame: Baseline, day 8 and day 15
Population: 1 participant in the sildenafil group was not able to tolerate 40 mg and did not reach the 15 day endpoint.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Sildenafil | Placebo Oral Tablet
Number analyzed (Participants) | 10 | 10
ratio
  Baseline | 0.10 [0.08 to 0.13] | 0.11 [0.09 to 0.12]
  Day 8 | 0.09 [0.06 to 0.15] | 0.12 [0.09 to 0.13]
  Day 15: number analyzed (Participants) | 9 | 10
  Day 15 | 0.06 [0.06 to 0.09] | 0.11 [0.08 to 0.15]

5. Other Pre Specified Outcome: Concentration of Serum Endothelin-1
Description: Mediator of vascular fibrosis. The normal reference is 1-2 pg/ml. Higher values indicate greater deviation from normal.
Time Frame: Baseline, day 8 and day 15
Population: 1 participant in the sildenafil group was not able to tolerate 40 mg and did not reach the 15 day endpoint.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Sildenafil | Placebo Oral Tablet
Number analyzed (Participants) | 10 | 10
pg/ml
  Baseline | 2.56 [2.35 to 2.78] | 2.78 [2.18 to 3.73]
  Day 8 | 2.27 [1.93 to 2.64] | 2.59 [2.10 to 3.93]
  Day 15: number analyzed (Participants) | 9 | 10
  Day 15 | 1.64 [1.62 to 2.09] | 2.66 [2.03 to 3.20]

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Sildenafil | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=10) | Placebo Oral Tablet (N=10)
Headache (Nervous system disorders) | 1 (1) | 0 (0) — 1 participant experienced a transient headache and could not tolerate 40 mg of sildenafil.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT03199612/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT03199612/ICF_001.pdf